CLINICAL TRIAL: NCT05550597
Title: Comparison of the Time to the First Rescue Analgesic Among Parturients Receiving Intrathecal Additive Fentanyl or Intrathecal Fentanyl With TAP Block or TAP Block Alone for Elective Cesarean Sections Under Hyperbaric Bupivacaine Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nepal Mediciti Hospital (Other)
Responsible Party: Principal Investigator, Bijay Rayamajhi, Anesthesia Resident, Nepal Mediciti Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022
Record Dates: First submitted 2022-09-13; First posted 2022-09-22 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Pain; Cesarean Section
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group F (Experimental): The intrathecal additive Fentanyl with hyperbaric bupivacaine
  Interventions: Drug: Fentanyl HCl
- Group FT (Experimental): The intrathecal additive of fentanyl with hyperbaric bupivacaine along with Ultrasound-guided TAP block
  Interventions: Drug: Fentanyl HCl; Drug: Bupivacaine 0.25% Injectable Solution
- Group T (Experimental): Hyperbaric bupivacaine along with Ultrasound-guided TAP block without the intrathecal addition of fentanyl
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Drug: Fentanyl HCl — Intrathecal additive Fentanyl with Hyperbaric Bupivacaine during Spinal Anesthesia
  Arms: Group F; Group FT
Drug: Bupivacaine 0.25% Injectable Solution — Intrathecal additive Fentanyl with Hyperbaric Bupivacaine during Spinal Anesthesia Ultrasound-guided Transversus Abdominal plane block using Bupivacaine 0.25% Injectable Solution
  Other Names: Intrathecal Fentanyl
  Arms: Group FT; Group T

SUMMARY:
The postoperative pain management after cesarean section under spinal anestheisa is done using various modalities. The commonly used regimens are systemic NSAIDs/Opioids, USG guided TAP block or Intrathecal additive Fentanyl or combined intrathecal fentanyl and USG guided TAP block.

Investigators aim to compare the postoperative analgesia in terms of time to the first rescue analgesic in parturients receiving intrathecal additive fentanyl only, or intrathecal fentanyl with USG guided TAP block or USG guided TAP block alone for elective CS done under hyperbaric bupivacaine spinal anesthesia.

DETAILED DESCRIPTION:
Investigators will enroll 93 parturients planned for elective CS under hyperbaric bupivacaine spinal anesthesia and allocate them into three groups comprising intrathecal additive fentanyl only, or intrathecal fentanyl with USG guided TAP block or USG guided TAP block alone.

The primary outcome will be time to the first rescue analgesics.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology(ASA) physical status II
* Able to read and understand the information sheet and to sign and date the consent form
* Scheduled for elective CS planned with Spinal anesthesia
* Gestational age > 37 weeks and < weeks assessed on the dating scale.

Exclusion Criteria:

* Complicated pregnancy; defined as having preeclampsia or placenta accreta,increta and percreta
* Opioid addiction or dependence
* Contraindications to TAP block( Ski infection, abdominal wall muscle defects)
* Allergy to any medications used in the study
* Case converted to General Anesthesia
* Cases who develop postoperative hemorrhage, amniotic fluid embolism

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
To compare the time to the first rescue analgesics | Time to first complain of pain with Numeric Rating scale(NRS) greater than or equal to 4 within first 24 hours
  The time from the arrival to Postoperative care Unit to first complain of pain with Numeric Rating scale(NRS) greater than or equal to 4 among the Parturients Receiving Intrathecal Additive Fentanyl or Intrathecal Fentanyl With TAP Block or TAP Block Alone for Elective Cesarean Sections Under Hyperbaric Bupivacaine Spinal Anesthesia

SECONDARY OUTCOMES:
Percentage of participants with treatment related side effects like pruritus, nausea and vomiting. | Time to first complain of pain with Numeric Rating scale(NRS) greater than or equal to 4 within first 24 hours
  To compare the side effects like pruritus, nausea and vomiting Among Parturients among the Parturients Receiving Intrathecal Additive Fentanyl or Intrathecal Fentanyl With TAP Block or TAP Block Alone for Elective Cesarean Sections Under Hyperbaric Bupivacaine Spinal Anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Bijay Rayamajhi, FCPS, Principal Investigator — Nepal Mediciti Hospital
Locations (1):
- Nepal Mediciti Hospital, Lalitpur, Nepal

IPD SHARING:
Plan to Share IPD: No